CLINICAL TRIAL: NCT01977027
Title: Strategies for Recovery of Dexterity Post Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left insitution
Sponsor: NYU Langone Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-03117; 1R01HD071978-01A1102617 (Other: National Institute of Child Health and Human Development); 1R01HD071978-01 (NIH)
Record Dates: First submitted 2013-08-23; First posted 2013-11-06 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Stroke With Hemiparesis
Keywords: Rehabilitation; Fingers; Grasp; Strength; Hand Function; Motor Function; Post Stroke; Brain Infraction; Biomechanis; Neuronal Plasticity; Weight-Bearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke & age-matched Controls (Other): Alternate Hand Training or Affected Hand Training:
  40 patients with stroke and 40 control subjects will participate over 7 visits. After completion of informed consent, subjects will undergo clinical assessments (Visit 1) which will involve testing for kinesthetic, visual, tactile and motor impairments and upper limb function. Visit 2, subjects will undergo no contrast MRI to identify lesion location. Healthy controls will not be imaged.
  Visits 3-7 will involve psychophysical experiments to test adaptation with short-term Alternate Hand Training and Affected Hand Training. During 5 visits the subjects will grasp and lift an instrumented grip device of different weights, textures and shapes while data is being collected via surface electrodes from, upper arm and back muscles.
  Interventions: Other: Alternate Hand Training or Affected Hand Training
- Phase 2 - Stroke ONLY (Other): Alternate Hand Training or Affected Hand Training:
  Subjects will be randomized into two groups one receiving Alternate Hand Training and the other receiving Affected Hand Training. The groups will be matched by age, gender, handedness, side of lesion, extent of motor impairment and lesion location. They will complete 17 Study visits.
  Visits 1 and 2 will involve clinical assessments and MRI. Visit 3. Pre-intervention assessments involving grasping and lifting objects of different weights, textures and shapes while fingertip forces, finger and arm movements. Muscle activity and performance is measured.
  Visits 4-15. Subjects will participate in 12 training visits for 1 hour a day, twice a week for 6 weeks.
  Visits 16-17. Recovery of hand function will be measured by repeating the pre-intervention clinical and grasping assessments (in 2 visits) immediately after 6-weeks of training, and another 6 weeks later.
  Interventions: Other: Alternate Hand Training or Affected Hand Training

INTERVENTIONS:
Other: Alternate Hand Training or Affected Hand Training — Participants will receive a training intervention with either the Alternate Hand Training Strategy, or Affected Hand Training alone.

SUMMARY:
Motor learning can be affected by the sensory difficulties that may be experienced as a result of a stroke. This study will help us better understand what kinds of sensory information can help with the re-learning of grasping with the affected hand despite the sensory difficulties produced by the stroke.

DETAILED DESCRIPTION:
The purpose of this study is to develop, refine and test the 'alternate hand training strategy' to facilitate adaptation, repetition and relearning to restore hand function after stroke. The three aims are: to restore adaptation (Aim 1), facilitate grasp efficiency and normal directional biases during repetition (Aim 2), and enhance the rate of learning to improve hand function and quality of life post stroke (Aim 3).

Hypotheses: We hypothesize that alternate hand training will increase the rate of learning and lead to greater improvement in hand function. The results will inform dosing of therapy for optimal relearning.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read/write in English
* Age > 18 yrs
* Radiologically verified stroke > 4 months old (3T structural MRI)
* Moderate arm motor impairment (Fugl-Meyer Scale < 60/66)
* Ability to reach, grasp and lift the test objects with the affected side as assessed by the PI
* Willingness to complete all clinical assessments and MRI, and comply with training protocols
* Ability to give informed consent and HIPPA certificationsPlease list all exclusion criteria for study:

Exclusion Criteria:

* Sensorimotor impairments in the unaffected hand
* Severe visual or sensory impairment, including neglect on the affected side
* Significant cognitive dysfunction (score < 24 on Folstein's Mini Mental Status Examination)
* Severe or unstable spasticity on treatment with Botulinum toxin or intrathecal baclofen
* Depression (Geriatric Depression Scale score <11)
* Major disability (modified Rankin Scale > 4)
* Previous neurological illness, complicated medical condition, or significant injury to either upper extremity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-08; Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
For Phase 1: Adaptation of fingertip forces and movements during grasping. | 6 weeks
  5 experiments will be performed over 7 visits to examine the best approach to retrain adaptation.
For Phase 2: Change in Hand function | 6 weeks
  Subjects will be randomized to Alternate Hand Training or Affected Hand Training arms and receive training twice a week for 6 weeks.

SECONDARY OUTCOMES:
Phase 2 - Maintenance of hand function | 6 weeks after end of training
  Recovery of hand function will be measured by repeating the pre-intervention clinical and grasping assessments 6-weeks after the end of training.

CONTACTS AND LOCATIONS:
Overall Officials: John R Rizzo, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States